CLINICAL TRIAL: NCT07005609
Title: Effects of Snakehead Fish as an Alternative High-Protein Food Source on Intrauterine Growth Restriction and Low Birth Weight Among Pregnant Women in Their Second and Third Trimesters Within Yogyakarta Province
Brief Title: Effects of Snakehead Fish on IUGR and LBW Among Second and Third Trimester Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Collaborators: National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other)
Responsible Party: Principal Investigator, Eugenius Phyowai Ganap, Principal Investigator, Gadjah Mada University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Snakehead Fish Meal
Record Dates: First submitted 2025-02-13; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-02

CONDITIONS: Pregnancy Related
Keywords: Snakehead fish prepared-meal; Intrauterine growth restriction; Low birth weight; Randomized controlled trial
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Snakehead Fish Meal Group (Experimental): Subjects in this treatment group received snakehead fish prepared-meal for about 3 months until delivery. Snakehead fish was provided at an amount of +-100 grams per serving.
  Interventions: Dietary Supplement: Snakehead fish meal
- Control Group (No Intervention): Subjects in this group did not receive snakehead fish intervention.

INTERVENTIONS:
Dietary Supplement: Snakehead fish meal — Subjects in the treatment group received snakehead fish meal daily for about 3 months until delivery. The meal contained carbohydrate, protein, vegetables and fruits. Snakehead fish was given +- 100 g per serving.
  Arms: Snakehead Fish Meal Group

SUMMARY:
This study uses a Randomized Controlled Trial (RCT) design, conducted on pregnant women in Yogyakarta Province, Indonesia. This study aims to observe the effects of snakehead fish prepared-meal intervention on fetal growth measurement and birth outcomes. The subjects were randomly divided into two groups (random allocation), the treatment and control groups. Subjects in the treatment group will be given supplementation of snakehead fish prepared-meal for lunch for 3 months daily, while subjects in the control group will not receive the intervention.

DETAILED DESCRIPTION:
Subjects in this study were divided into two groups; treatment group, who were given snakehead fish prepared-meal for lunch everyday, and control group who were not given any supplementation.All participants have already agreed to join this study by signing the informed consent at the beginning of the study.

Snakehead fish meal contained carbohydrate, protein (from snakehead fish), vegetables and fruit. The daily intake of snakehead fish meal were noted in the food record form independently by the subjects in the treatment group and would be reported periodically to the researcher. Snakehead fish meal were given for about 3 months or until the mother deliver the baby.

All participants in both group were examined once a month using 2D ultrasonography to measured fetal growth. After the baby was born, baby's birth weigth and birth length data were obtained through the mother and baby's health book.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 28 years
2. In the 2nd and 3rd trimesters
3. Middle to lower economic status

Exclusion Criteria:

1. Anemia
2. Preeclampsia
3. Multiple gestational pregnancy
4. Allergies to fish

Max Age: 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Subjects in this study were pregnant women in the second and third trimesters.
Enrollment: 56 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Snakehead fish intake | Snakehead fish intake were noted using food record every day for about 3 months.
  The daily intake of snakehead fish meal of the treatment group were measured using Food Intake Record form. The intake of the meal were categorized as finished (100%), 3/4 (75%), 1/2 (50%), 1/4 (25%), not eaten at all (0%). The higher the intake, the better the acceptability of the snakehead fish meal.
Estimated Fetal Weight (EFW) | Estimated fetal weight was measured 3 times using 2D-Ultrasound once every 4 weeks, around week 1, week 5, and week 9 of the study.
  Primary outcomes measured in this study were fetal growth. One of the fetal growth indicator was estimated fetal weight (EFW), reported in grams.
Femur length (FL) | Femur length was measured 3 times using 2D-Ultrasound once every 4 weeks, around week 1, week 5, and week 9 of the study.
  Femur length was also one of the fetal growth indicator measured in this study. It was noted in centimeters.
Biparietal diameter (BPD) | Biparietal diamter was measured 3 times using 2D-Ultrasound once every 4 weeks, around week 1, week 5, and week 9 of the study.
  Biparietal diameter was also measured along with EFW and FL, reported in centimeters.
Head circumference (HC) | Head circumference was measured 3 times using 2D-Ultrasound once every 4 weeks, around week 1, week 5, and week 9 of the study.
  Head circumference of the baby was also measured in this study. It is noted in centimeters.
Abdominal circumference (AC) | Abdominal circumference was measured 3 times using 2D-Ultrasound once every 4 weeks, around week 1, week 5, and week 9 of the study.
  Abdominal circumference was another fetal growth indicator that also be measured during this study, and was reported in centimeters.
Birth weight | at the end of the study completion (after the baby is born), after an average of 3 months.
  Baby's birth weight data were collected from the mother and child's health book.
Birth length | at the end of the study completion (after the baby is born), after an average of 3 months.
  Baby's birth length data were collected from the mother and child's health book.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenius P Ganap, PhD, Principal Investigator — Department of Obstetric and Gynecology, Faculty of Medicine, Public Health and Nursing, Universitas Gadjah Mada, Yogyakarta, Indonesia
Locations (1):
- Obstetric and Gynecology Department, Faculty of Medicine, Public Health, and Nursing, Universitas Gadjah Mada, Sleman, Special Region of Yogyakarta, Indonesia